CLINICAL TRIAL: NCT03533465
Title: Understanding the Role of Sleep in Complicated Grief: A Pilot Study
Brief Title: Understanding the Role of Sleep in Complicated Grief
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to funding limitations
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-00003
Record Dates: First submitted 2018-04-18; First posted 2018-05-23 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Sleep; Grief

STUDY DESIGN:
Intervention Model Description: The first aim of this study will involve a comparison of baseline psychiatric symptoms and subjective and objective measures of sleep, with specific attention to REM, in adults with CG compared to 25 healthy controls. 10 of these adults with CG who complete AIM 1 will participate in Complicated Grief Treatment (CGT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Complicated Grief Treatment (CGT) (Experimental): 10 adults with CG who successfully completed Aim 1 and will also participate in open complicated grief treatment (CGT), during which they will complete additional subjective and objective sleep assessments.
  Interventions: Behavioral: Complicated Grief Therapy (CGT)

INTERVENTIONS:
Behavioral: Complicated Grief Therapy (CGT) — CGT is an evidence based 16 session targeted grief therapy delivered in individual one hour weekly sessions. Treatment will end at 16 sessions (offered over the course of 20 weeks)

SUMMARY:
The purpose of this study is to learn more about the causes of Complicated Grief (CG) in those who experience the loss of a loved one. This study aims at learning more about the sleep patterns and emotions in participants with CG as compared to those who have lost a loved one but do not have CG.

This study will consist of two aims:

Aim 1: Approximately 10 complicated grief (CG) patients and 10 controls (without a current psychiatric diagnosis) will complete a 3-day home polysomnography (PSG) sleep assessment in addition to several self-report sleep and psychiatric measures.

Aim 2: Approximately 10 CG patients (subsample from Aim 1) will complete 16 weekly sessions of complicated grief therapy (CGT) in addition to completion of repeated PSG assessments and self-report sleep and psychiatric measures.

ELIGIBILITY:
Inclusion Criteria:

* Bereaved due to death of a loved one >= 6 months prior (for both CG and control groups)
* For CG participants: grief is primary psychiatric problem with ICG >= 30 (threshold symptoms; for CG group only). Controls will be free of current psychiatric disorders with the exception of specific phobia.
* Normal or corrected vision

Exclusion Criteria:

* Psychiatric or sleep medications in the past 4 weeks (past 6 weeks for fluoxetine)
* Concurrent grief or exposure based therapy
* Lifetime bipolar, psychosis, significant neurological disorders
* Past 6 months of alcohol/substance use disorder
* Unstable medical illness
* Serious safety concerns of suicide or homicide
* Pregnant or nursing
* Overnight shift work
* > 4 caffeinated or > 11 alcoholic beverages per week
* Screening reveals OSA defined as an apnea hypopnea index with 4% desaturation (AHI4%) ≥15 or an AHI4% ≥ with an Epworth >10

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2019-03-25 (Actual); Study Completion 2019-03-25 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression Scales | 16 Weeks
  Measure of Clinical Improvement and Severity of illness on a scale of 1-7; 1 being "Very Much Improved"; 7 being Very Much Worse

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Simon, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States